CLINICAL TRIAL: NCT03365700
Title: Cryoballon Versus Conventional Radiofrequency Ablation for Persistent Atrial Fibrillation With AF Duration < 2 Years: the IRON-ICE Trial
Brief Title: Cryoballon Versus Radiofrequency Ablation for Persistent Atrial Fibrillation
Acronym: IRON-ICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luigi Sacco University Hospital (Other)
Collaborators: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Giovanni B Forleo, Section Head Electrophysiology and Cardiac Pacing., Luigi Sacco University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRON2017
Record Dates: First submitted 2017-11-17; First posted 2017-12-07 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Persistent atrial fibrillation; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryoballoon ablation (Active Comparator): Cryoballoon pulmonary vein isolation with the Arctic Front Advance® System or any future development generations of this product line.
  Interventions: Procedure: Cryoballoon ablation
- Radiofrequency Ablation (Active Comparator): Contact force-sensing radiofrequency left atrial ablation with 3D mapping system.
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Radiofrequency Ablation — Left atrial catheter ablation with pulmonary vein antrum isolation documented by a circular mapping catheter.
  Other Names: Pulmonary vein isolation
  Arms: Radiofrequency Ablation
Procedure: Cryoballoon ablation — Cryoballoon pulmonary vein isolation with the Arctic Front Advance® System or any future development generations of this product line. Additional substrate modification is allowed with the catheter type assigned at the index procedure.
  Other Names: Pulmonary vein isolation
  Arms: Cryoballoon ablation

SUMMARY:
A randomized trial has recently demonstrated non-inferiority of cryoballoon vs. radiofrequency (RF) catheter ablation in patients with drug-refractory paroxysmal atrial fibrillation (AF). There is a growing amount of evidence suggesting that Cryoballoon ablation is highly effective also in non-paroxysmal atrial fibrillation.

The IRON-ICE trial will evaluate the effect of Cryoballoon AF ablation in patients with short-term persistent AF.

ELIGIBILITY:
Inclusion Criteria:

1. Candidates for AF ablation based on AF that is symptomatic and refractory to at least one antiarrhythmic medication.
2. Patients presenting with Persistent AF with AF duration < 2 years scheduled to undergo a PVAI procedure
3. Age range of 18 - 85 years
4. Patients with already implanted devices with AF detection capabilities (for clinical indications): ILR implanted in the same hospital stay or within 6 months before the ablation or patients with an dual chamber PM, ICD or CRTD and an existing functional atrial lead.
5. Patients must be able and willing to provide written informed consent to participate in the clinical trial.

Exclusion Criteria:

* Congenital heart disease, age younger than 18 years, significant valve disease, LA size >55 mm, and severe heart failure (ejection fraction < 30% and/or New York Heart Association class IV).
* Presence of a mechanical prosthetic valve.
* Secondary causes of atrial fibrillation
* Documented intra-atrial thrombus or another abnormality which precludes catheter introduction.
* Social factors that would preclude follow up or make compliance difficult.-
* Patients who are or may potentially be pregnant Previous left atrial catheter ablation or MAZE procedure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial tachycardia/fibrillation | 12 months
  Freedom from atrial tachycardia/fibrillation within 12 months after CA. Arrhythmias had to last 30 seconds or more to be considered present.

SECONDARY OUTCOMES:
Number of AF episodes recorded. | 12 months
Duration of AF episodes recorded. | 12 months
Length of postoperative hospital stay. | 1 month
Total procedural time. | 1 day
Fluoroscopy time | 1 day
Left atrial instrumentation time | 1 day
  total time during which there are catheters in the LA
Hospitalizations after discharge. | 12 months
  number of hospitalizations after discharge
Procedure-related complications | 1 week
  Complications: cerebrovascular (thromboembolic or hemorrhagic), cardiovascular (cardiac perforation, tamponade) or gastrointestinal.
Incidence of cerebrovascular events from the time of the operation up to 90 days. | 90 Days
Long-term success | 36 months
  freedom from AF/AFL/AT recurrences following the 3-month blanking period within 36-month follow-up from the date of the ablation procedure in the absence of Class I and III antiarrhythmic drug therapy.
Freedom from clinical or stroke-relevant AF/AFL/AT. | 12 months
  Freedom from AF/AFL/AT with duration cutoff > 1 hour
Freedom from persistent AF/AFL/AT (duration cutoff of 7 days) | 12 months
  Freedom from AF/AFL/AT with duration cutoff > 7 days
Regression from persistent to non-paroxysmal atrial fibrillation | 12 months
  Patients converted into paroxysmal forms of AF.
Significant reduction in AF burden | 12 months
  >75% reduction from pre- to postablation and/or total postablation burden <12%
Low daily AF burden | 12 months
  Patients with AF burden less than 1%- 2%
Death from any cause | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Tondo, MD, PhD, Principal Investigator — Heart Rhythm Center at Monzino Cardiac Center, IRCCS.
Locations (3):
- Italy (3):
  - Azienda Ospedaliera - Polo Universitario - "Luigi Sacco", Milan
  - Heart Rhythm Center at Monzino Cardiac Center, IRCCS., Milan
  - Istituto Clinico S. Ambrogio, Milan

REFERENCES:
- [Result] Kuck KH, Furnkranz A, Chun KR, Metzner A, Ouyang F, Schluter M, Elvan A, Lim HW, Kueffer FJ, Arentz T, Albenque JP, Tondo C, Kuhne M, Sticherling C, Brugada J; FIRE AND ICE Investigators. Cryoballoon or radiofrequency ablation for symptomatic paroxysmal atrial fibrillation: reintervention, rehospitalization, and quality-of-life outcomes in the FIRE AND ICE trial. Eur Heart J. 2016 Oct 7;37(38):2858-2865. doi: 10.1093/eurheartj/ehw285. Epub 2016 Jul 5. PMID 27381589
- [Result] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964